CLINICAL TRIAL: NCT05075642
Title: A Multicentre Observational Study for the Evaluation in Clinical Practice of the Initial Diagnostic-therapeutic Path of Urinary Disorders in Multiple Sclerosis
Brief Title: Multicenter Observational Study for the Evaluation in Clinical Practice of Urinary Disorders in Multiple Sclerosis
Acronym: MUSA
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: ASP 7 Ragusa (Other)
Responsible Party: Principal Investigator, Carmela Leone, Principal Investigator, ASP 7 Ragusa
Other Study IDs: E - 0027793
Record Dates: First submitted 2021-09-19; First posted 2021-10-13 (Actual); Last update posted 2021-10-13 (Actual); Status verified 2021-09

CONDITIONS: Multiple Sclerosis; Urinary Bladder, Neurogenic
Keywords: Patient global impression of improvement; management; treatment; low urinary tract symptoms; diagnostic tools; prevalence
MeSH Terms: conditions — Multiple Sclerosis; Urinary Bladder, Neurogenic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Initial management of the urinary disorder/s identified during the screening phase — Intervention can be defined as the initial management of the LUTS identified during the screening phase; management lasts at least three months. As observation of routine clinical practice, no specific intervention is included, but any counseling/drug/rehabilitation included as first line management.

SUMMARY:
The major part of people with multiple sclerosis (pwMS) experiences Low Urinary Tract Symptoms (LUTS) secondary to neurogenic Low Urinary Tract Dysfunctions (n-LUTDs) during the course of MS, reaching almost 100% after about 10 years. N-LUTDs represent an important issue for pwMS, especially for their negative impact on Quality of Life (QoL), as they are mainly youngs in the prime of their life. Moreover n-LUTDs can lead to serious complications on the urinary tract as infections or renal failure. Therefore, the neurologist in daily clinical practice must intercept the possible presence of LUTS as soon as possible so that he can promptly initiate optimal management. To do this, it is essential to provide neurologists with validated, reproducible and sensitive tools that are, above all, easy to use in an outpatient setting. Our clinical research seeks, for the first time, to show whether pwMS get any improvement after the initial LUTS management, whether this improvement, if any, is related to the professional figure takes care about LUTS (neurologist vs urologist) and if there is an objective improvement of voiding performances on standardized measures.

DETAILED DESCRIPTION:
The investigators will conduct a multicenter observational no-profit study to investigate the impact of Low Urinary Tract Symptoms (LUTS) management on subjective measure of patient global impression of improvement.

Initial management of LUTS in MS should address both voiding and storage deficiency symptoms and is determined by the severity of symptoms and the risk of developing upper urinary tract damage. First-line treatments include behavioral / physical ones, such as rehabilitation of the pelvic floor, and pharmacological ones (antimuscarinics, alpha-lytics, beta3 agonists); second-line treatments are represented by intradetrusorial (or intrasphinteric) injection of botulinum toxin and by non-invasive (percutaneous and transcutaneous tibial nerve stimulation) and invasive (sacral neuromodulation) neuromodulation techniques; third-line treatments consist of surgical approaches. According to the various consensus and recommendations available for MS, the initial approach in most cases should be the prerogative of the neurologist, while the neurourologist should intervene when the initial treatment has been ineffective or there are pathologies of the urinary tract that require a non-postponable specialist evaluation.

As regards the effectiveness of any initial management of LUTS in pcSM, there are, to the best of our knowledge, no studies in the literature that have analyzed the phenomenon, both in terms of subjective perception of clinical improvement and in objective terms of objective improved "voiding performance".

This study was developed with the primary intention of measuring, through the observation of real clinical practice, the presence and extent of improvement (through the PGI-I scale) of the subject with LUTS after at least three months of any type of initial management. A subgroup analysis will help us to assess whether the neurologist's management of LUTS is different from that of the urologist in terms of perceived improvement.

A patient reported outcome assessing quality of life (Qualiveen-SF), a three-day frequency / volume chart, and post-voiding residual volume (PVR) will be used as secondary outcomes to reveal the effectiveness of the two approaches on quality of life and data objective measures of urinary disorders.

The study also aims to 1) evaluate the prevalence of LUTS through a new diagnostic algorithm that consists of two questionnaires (the Urinary Bothersome Questionnaire-MS and the Actionable Bladder Symptoms Screening Tool-ABSST) and an objective measure of voiding dysfunction-the PVR and 2) analyze the influence of the more common risk factors on the presence of LUTS as thus diagnosed.

ELIGIBILITY:
Inclusion Criteria:

* People with MS (relapsing-remitting, secondary progressive, primary progressive phenotype) or clinically isolated demyelinating disease syndrome-CIS) according to McDonald's 2001 criteria, consecutively afferent to the outpatient clinic or hospitalized after study approval by the ethics committee.

They:

* have never been previously evaluated and/or treated for LUTS secondary to MS;
* are between 18 and 80 years old;
* have given written consent to study part.

Exclusion Criteria:

* analphabetism;
* severe cognitive impairment;
* severe psychiatric pathologies;
* EDSS> 7;
* clinical relapse of MS within the previous 30 days;
* history of urinary fevers > 2 in the last 6 months or > 3 in the last year;
* indwelling catheter;
* renal failure (creatinine> 1.2 mg / dL);
* presence of hydronephrosis, mono or bilateral vesicoureteral reflux;
* presence of urinary stones;
* history of urological surgery, neoplasms of the urogenital system and / or pelvic radiotherapy;
* therapy/treatment for LUTS secondary to MS or other diseases.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: For this study, a total of 214 persons with MS will be recruited. They will be recruited from the patients consecutively will attend the clinic or will be admitted to the participating Multiple Sclerosis Center, after approval of the study by the respective ethics committee
Sampling Method: Probability Sample
Enrollment: 214 (Estimated)
Dates: Start 2021-11 (Estimated); Primary Completion 2023-05 (Estimated); Study Completion 2023-07 (Estimated)

PRIMARY OUTCOMES:
Patient global impression of Improvement (PGI-I) questionnaire | at the end-of-study visit named Visit 2, corresponding at week 12-16 from Visit 1, that is the management start-up visit
  In participants with recorded LUTS, it will be measured the subjective impression of improvement after at least three months of stable urinary disorder management, by means of the PGI-I questionnaire. The PGI-I is a 1-item questionnaire designed to assess the patient's impression of change with values ranging from 1 to 7; higher scores mean a worse outcome. Patient is required to "Check the one number that best describes how you feel now" by entering his answer on a 7-point scale scored as: (1) "very much better," (2) "much better," (3) "a little better," (4) "no change," (5) "a little worse," (6) "much worse," or (7) "very much worse." For this study, investigators will evaluated as primary outcome measure "the percentage of patient gave a response to PGI-I equal to or less than 2".

SECONDARY OUTCOMES:
Qualiveen-Short Form (SF) questionnaire | at the end of screening period named Visit 0, and at Visit 2 (weeks 12-16 from Visit 1, that is the management start-up visit)
  In participants with recorded LUTS, it will be measured the patient reported urinary-related quality of life by means of the Qualiveen-Short Form (SF) questionnaire. It's a specific health related quality of life (HRQOL) with questionnaire for urinary disorders in patients with neurological conditions, such as Multiple Sclerosis.
  The Qualiveen-SF is an 8-items questionnaire. Response options are framed as 5-point Likert-type scales with 0 indicating no impact of urinary problems on HRQOL and 4 indicating a high adverse impact of urinary difficulty on HRQOL. Qualiveen domain scores are calculated as an average of the scores on items in that domain and, thus, the range is 0 to 4 with an overall score representing the mean of the 4 domains, which also ranges from 0 to 4. Higher scores mean worse outcome.
  For this study investigators will evaluated whether three-months (max 4 months) of urinary disorder stable management may change HRQOL in terms of Qualiveen-SF scores.
Post-void residual volume (PVR) assessment | at visit 0 and Visit 2 (weeks 12-16 from Visit 1, that is the management start-up visit)
  The post-void residual volume (PVR) measured in ml is the urine volume remaining in bladder after a physiological micturition. It will be measured by ultrasound scans and calculated by the radiologist subtracting post-void bladder volume from pre-void bladder volume.
  For this study, the investigators will evaluate whether three months (max 4 months) of urinary disorder stable management may change the amount of PVR.
  Lower volume values mean better outcome.
Micturitions' frequency and episodes of urgency/incontinence at three days frequency/volume chart | at visit 0 and Visit 2 (weeks 12-16 from Visit 1, that is the management start-up visit)
  In participants with recorded LUTS, it will be measured the number of daily micturitions and episodes of urgency or incontinence signed on a three days frequency/volume chart. Frequency/volume chart is a brief diary where patients are asked to record for three days how many times they urinate and the volume of each micturition; they are also asked to record each episode of urinary urgency and incontinence. Higher numbers mean worse outcome.
  As secondary outcome, it will be evaluated whether three months (max 4 months) of urinary disorder stable management may change the numbers of micturitions and numbers of urinary urgency and/or incontinence.

OTHER OUTCOMES:
Prevalence of LUTS | at Visit 0 (screening visit)
  Considering all participants underwent screening visit, it will be estimated the prevalence of Low Urinary Tract Symptoms (LUTS); a new diagnostic screening model consisting of the Urinary Bothersome Questionnaire for Multiple Sclerosis (UBQ-MS), the Actionable Bladder Symptoms Screening Tool (ABSST) questionnaire and the PVR volume is used; LUTS is defined by the presence of at least one diagnostic tool with abnormal finding: UBQ-MS score at least 1, ABSST at least 3, PVR at least 100 ml or more than 30% of pre-void assessed volume.
Demographic, Clinical and instrumental characteristics | at visit 0 (screening visit)
  Evaluating the presence of demographic (age, sex, BMI), clinical (disease duration, phenotype, Expanded Disease Status Scale, spinal lesions and their location, therapy, comorbidities) and instrumental factors (urinalysis with urine culture, radiological imaging, number of urinations and urgency-frequency episodes with frequency / volume chart) predictive of the type of urinary disorders reported.
Patient global impression of Improvement (PGI-I) questionnaire, Qualiveen-Short Form questionnaire, Post-void residual volume (PVR) amount, Micturitions' frequency and episodes of urgency/incontinence at three days frequency/volume chart | at visit 0 (screening visit) and visit 2 (weeks 12-16 from Visit 1, that is the management start-up visit)
  Finally, by means of a subgroup analysis, the investigators will evaluate whether enrolled participants managed by neurologists or by urologists show any difference in scores of Patient global impression of Improvement (PGI-I) questionnaire, Qualiveen-Short Form questionnaire, Post-void residual volume (PVR) assessment, Micturitions' frequency and episodes of urgency/incontinence at three days frequency/volume chart.
  According to the specific MS center clinical practice, patients with MS may be managed by the neurologist or by the urologist by the urologist to whom they will be referred.

CONTACTS AND LOCATIONS:
Overall Officials: Carmela Leone, MD, Principal Investigator — Multiple Sclerosis Center of ASP7 Ragusa; Antonello Giordano, MD, Study Director — Multiple Sclerosis Center of ASP7 Ragusa
Locations (1):
- Multiple Sclerosis Center of ASP 7 Ragusa, Vittoria, Ragusa, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] de Seze M, Ruffion A, Denys P, Joseph PA, Perrouin-Verbe B; GENULF. The neurogenic bladder in multiple sclerosis: review of the literature and proposal of management guidelines. Mult Scler. 2007 Aug;13(7):915-28. doi: 10.1177/1352458506075651. Epub 2007 Mar 15. PMID 17881401
- [Result] Panicker JN, Fowler CJ, Kessler TM. Lower urinary tract dysfunction in the neurological patient: clinical assessment and management. Lancet Neurol. 2015 Jul;14(7):720-32. doi: 10.1016/S1474-4422(15)00070-8. PMID 26067125
- [Result] Khalaf KM, Coyne KS, Globe DR, Malone DC, Armstrong EP, Patel V, Burks J. The impact of lower urinary tract symptoms on health-related quality of life among patients with multiple sclerosis. Neurourol Urodyn. 2016 Jan;35(1):48-54. doi: 10.1002/nau.22670. Epub 2014 Oct 18. PMID 25327401
- [Result] Musco S, Padilla-Fernandez B, Del Popolo G, Bonifazi M, Blok BFM, Groen J, 't Hoen L, Pannek J, Bonzon J, Kessler TM, Schneider MP, Gross T, Karsenty G, Phe V, Hamid R, Ecclestone H, Castro-Diaz D. Value of urodynamic findings in predicting upper urinary tract damage in neuro-urological patients: A systematic review. Neurourol Urodyn. 2018 Jun;37(5):1522-1540. doi: 10.1002/nau.23501. Epub 2018 Feb 2. PMID 29392753
- [Result] Groen J, Pannek J, Castro Diaz D, Del Popolo G, Gross T, Hamid R, Karsenty G, Kessler TM, Schneider M, 't Hoen L, Blok B. Summary of European Association of Urology (EAU) Guidelines on Neuro-Urology. Eur Urol. 2016 Feb;69(2):324-33. doi: 10.1016/j.eururo.2015.07.071. Epub 2015 Aug 22. PMID 26304502
- [Result] Litwiller SE, Frohman EM, Zimmern PE. Multiple sclerosis and the urologist. J Urol. 1999 Mar;161(3):743-57. PMID 10022678
- [Result] Grasso MG, Pozzilli C, Anzini A, Salvetti M, Bastianello S, Fieschi C. Relationship between bladder dysfunction and brain MRI in multiple sclerosis. Funct Neurol. 1991 Jul-Sep;6(3):289-92. PMID 1743544
- [Result] Fowler CJ, Griffiths D, de Groat WC. The neural control of micturition. Nat Rev Neurosci. 2008 Jun;9(6):453-66. doi: 10.1038/nrn2401. PMID 18490916
- [Result] Griffiths D, Tadic SD. Bladder control, urgency, and urge incontinence: evidence from functional brain imaging. Neurourol Urodyn. 2008;27(6):466-74. doi: 10.1002/nau.20549. PMID 18092336
- [Result] Ghezzi A, Carone R, Del Popolo G, Amato MP, Bertolotto A, Comola M, Del Carro U, Di Benedetto P, Giannantoni A, Lopes de Carvalho ML, Montanari E, Patti F, Protti A, Rasia S, Salonia A, Scandellari C, Sperli F, Spinelli M, Solaro C, Uccelli A, Zaffaroni M, Zipoli V; Multiple Sclerosis Study Group, Italian Society of Neurology. Recommendations for the management of urinary disorders in multiple sclerosis: a consensus of the Italian Multiple Sclerosis Study Group. Neurol Sci. 2011 Dec;32(6):1223-31. doi: 10.1007/s10072-011-0794-y. PMID 21948057
- [Result] De Ridder D, Van Der Aa F, Debruyne J, D'hooghe MB, Dubois B, Guillaume D, Heerings M, Ilsbroukx S, Medaer R, Nagels G, Seeldrayers P, Van Landegem W, Willekens B, Zicot AF. Consensus guidelines on the neurologist's role in the management of neurogenic lower urinary tract dysfunction in multiple sclerosis. Clin Neurol Neurosurg. 2013 Oct;115(10):2033-40. doi: 10.1016/j.clineuro.2013.06.018. Epub 2013 Jul 20. PMID 23880016
- [Result] Medina-Polo J, Adot JM, Allue M, Arlandis S, Blasco P, Casanova B, Matias-Guiu J, Madurga B, Meza-Murillo ER, Muller-Arteaga C, Rodriguez-Acevedo B, Vara J, Zubiaur MC, Lopez-Fando L. Consensus document on the multidisciplinary management of neurogenic lower urinary tract dysfunction in patients with multiple sclerosis. Neurourol Urodyn. 2020 Feb;39(2):762-770. doi: 10.1002/nau.24276. Epub 2020 Jan 15. PMID 31943361
- [Result] Bates D, Burks J, Globe D, Signori M, Hudgens S, Denys P, Macdiarmid S, Nitti V, Odderson I, Ross AP, Chancellor M. Development of a short form and scoring algorithm from the validated actionable bladder symptom screening tool. BMC Neurol. 2013 Jul 9;13:78. doi: 10.1186/1471-2377-13-78. PMID 23837535
- [Result] Burks J, Chancellor M, Bates D, Denys P, Macdiarmid S, Nitti V, Globe D, Signori M, Hudgens S, Odderson I, Panicker J, Ross AP. Development and validation of the actionable bladder symptom screening tool for multiple sclerosis patients. Int J MS Care. 2013 Winter;15(4):182-92. doi: 10.7224/1537-2073.2012-049. PMID 24453782
- [Result] Denys P, Phe V, Even A, Chartier-Kastler E. Therapeutic strategies of urinary disorders in MS. Practice and algorithms. Ann Phys Rehabil Med. 2014 Jul;57(5):297-301. doi: 10.1016/j.rehab.2014.05.003. Epub 2014 Jun 4. PMID 24958444
- [Result] Tsang B, Stothers L, Macnab A, Lazare D, Nigro M. A systematic review and comparison of questionnaires in the management of spinal cord injury, multiple sclerosis and the neurogenic bladder. Neurourol Urodyn. 2016 Mar;35(3):354-64. doi: 10.1002/nau.22720. Epub 2015 Jan 25. PMID 25620137
- [Result] Welk B, Morrow S, Madarasz W, Baverstock R, Macnab J, Sequeira K. The validity and reliability of the neurogenic bladder symptom score. J Urol. 2014 Aug;192(2):452-7. doi: 10.1016/j.juro.2014.01.027. Epub 2014 Feb 8. PMID 24518764
- [Result] Al Dandan HB, Coote S, McClurg D. Prevalence of Lower Urinary Tract Symptoms in People with Multiple Sclerosis: A Systematic Review and Meta-analysis. Int J MS Care. 2020 Mar-Apr;22(2):91-99. doi: 10.7224/1537-2073.2019-030. PMID 32410904
- [Result] Amarenco G, Chartier-Kastler E, Denys P, Jean JL, de Seze M, Lubetzski C. First-line urological evaluation in multiple sclerosis: validation of a specific decision-making algorithm. Mult Scler. 2013 Dec;19(14):1931-7. doi: 10.1177/1352458513489758. Epub 2013 May 22. PMID 23698129
- [Result] Bonniaud V, Bryant D, Parratte B, Guyatt G. Qualiveen, a urinary-disorder specific instrument: 0.5 corresponds to the minimal important difference. J Clin Epidemiol. 2008 May;61(5):505-10. doi: 10.1016/j.jclinepi.2007.06.008. Epub 2008 Jan 7. PMID 18394545
- [Result] Bonniaud V, Bryant D, Parratte B, Guyatt G. Development and validation of the short form of a urinary quality of life questionnaire: SF-Qualiveen. J Urol. 2008 Dec;180(6):2592-8. doi: 10.1016/j.juro.2008.08.016. Epub 2008 Oct 31. PMID 18950816
- [Result] Domurath B, Kurze I, Kirschner-Hermanns R, Kaufmann A, Feneberg W, Schmidt P, Henze T, Flachenecker P, Brandt A, Vance WN, Beck J, Vonthien M, Ratering K; MS Consensus Group. Neurourological assessment in people with multiple sclerosis (MS): a new evaluated algorithm. Mult Scler Relat Disord. 2020 Sep;44:102248. doi: 10.1016/j.msard.2020.102248. Epub 2020 May 30. PMID 32562907
- [Result] Li V, Panicker JN, Haslam C, Chataway J. Use of a symptom-based questionnaire to screen for the presence of significant voiding dysfunction in patients with multiple sclerosis and lower urinary tract symptoms: a pilot study. J Neurol. 2020 Dec;267(12):3683-3688. doi: 10.1007/s00415-020-10068-2. Epub 2020 Jul 16. PMID 32671529
- [Result] Ghezzi A, Mutta E, Bianchi F, Bonavita S, Buttari F, Caramma A, Cavarretta R, Centonze D, Coghe GC, Coniglio G, Del Carro U, Ferro MT, Marrosu MG, Patti F, Rovaris M, Sparaco M, Simone I, Tortorella C, Bergamaschi R. Diagnostic tools for assessment of urinary dysfunction in MS patients without urinary disturbances. Neurol Sci. 2016 Mar;37(3):437-42. doi: 10.1007/s10072-015-2415-7. Epub 2015 Nov 27. PMID 26613723
- [Result] Monti Bragadin M, Motta R, Messmer Uccelli M, Tacchino A, Ponzio M, Podda J, Konrad G, Rinaldi S, Della Cava M, Battaglia MA, Brichetto G. Lower urinary tract dysfunction in patients with multiple sclerosis: A post-void residual analysis of 501 cases. Mult Scler Relat Disord. 2020 Oct;45:102378. doi: 10.1016/j.msard.2020.102378. Epub 2020 Jul 5. PMID 32683303
- [Result] Yalcin I, Bump RC. Validation of two global impression questionnaires for incontinence. Am J Obstet Gynecol. 2003 Jul;189(1):98-101. doi: 10.1067/mob.2003.379. PMID 12861145
- [Result] Bjelic-Radisic V, Ulrich D, Hinterholzer S, Reinstadler E, Geiss I, Aigmueller T, Tamussino K, Greimel E, Trutnovsky G; Austrian Urogynecology Working Group. Psychometric properties and validation of two global impression questionnaires (PGI-S, PGI-I) for stress incontinence in a German-speaking female population. Neurourol Urodyn. 2018 Apr;37(4):1365-1371. doi: 10.1002/nau.23447. Epub 2017 Nov 11. PMID 29130524
- [Result] Viktrup L, Hayes RP, Wang P, Shen W. Construct validation of patient global impression of severity (PGI-S) and improvement (PGI-I) questionnaires in the treatment of men with lower urinary tract symptoms secondary to benign prostatic hyperplasia. BMC Urol. 2012 Nov 7;12:30. doi: 10.1186/1471-2490-12-30. PMID 23134716
- [Result] Twiss CO, Fischer MC, Nitti VW. Comparison between reduction in 24-hour pad weight, International Consultation on Incontinence-Short Form (ICIQ-SF) score, International Prostate Symptom Score (IPSS), and Post-Operative Patient Global Impression of Improvement (PGI-I) score in patient evaluation after male perineal sling. Neurourol Urodyn. 2007;26(1):8-13. doi: 10.1002/nau.20333. PMID 17016797
- [Result] McDonald WI, Compston A, Edan G, Goodkin D, Hartung HP, Lublin FD, McFarland HF, Paty DW, Polman CH, Reingold SC, Sandberg-Wollheim M, Sibley W, Thompson A, van den Noort S, Weinshenker BY, Wolinsky JS. Recommended diagnostic criteria for multiple sclerosis: guidelines from the International Panel on the diagnosis of multiple sclerosis. Ann Neurol. 2001 Jul;50(1):121-7. doi: 10.1002/ana.1032. PMID 11456302
- [Result] Polman CH, Reingold SC, Banwell B, Clanet M, Cohen JA, Filippi M, Fujihara K, Havrdova E, Hutchinson M, Kappos L, Lublin FD, Montalban X, O'Connor P, Sandberg-Wollheim M, Thompson AJ, Waubant E, Weinshenker B, Wolinsky JS. Diagnostic criteria for multiple sclerosis: 2010 revisions to the McDonald criteria. Ann Neurol. 2011 Feb;69(2):292-302. doi: 10.1002/ana.22366. PMID 21387374
- [Result] Bates P, Bradley WE, Glen E, Melchior H, Rowan D, Sterling A, Hald T. The standardization of terminology of lower urinary tract function. Eur Urol. 1976;2(6):274-6. doi: 10.1159/000472029. PMID 1036165